CLINICAL TRIAL: NCT02819986
Title: Effectiveness and Feasibility of Using the Progressive Goal Attainment Program in Anxiety and Mood Disorders
Brief Title: Effectiveness of Using the Progressive Goal Attainment Program in Anxiety and Mood Disorders
Acronym: PGAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Tanja Colonerus, Priniciple Investigator, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1784
Record Dates: First submitted 2016-06-20; First posted 2016-06-30 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Anxiety; Mood Disorder
Keywords: occupational functioning; Worries; Pain; Disability
MeSH Terms: conditions — Anxiety Disorders; Mood Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Progressive Goal Attainment Program (Experimental): 10 one hour weekly therapy sessions focused on behavioural interventions
  Interventions: Behavioral: Progressive Goal Attainment Program

INTERVENTIONS:
Behavioral: Progressive Goal Attainment Program — Behavioural intervention that consists of 10 one hour weekly therapy sessions that focus on goal setting, challenging thoughts about return to work, problem solving, behavioural activation, and resuming occupational roles.
  Other Names: PGAP

SUMMARY:
The purpose of the present study is to determine the effectiveness and feasibility of the Progressive Goal Attainment Program (PGAP) with individuals with anxiety and mood disorders. PGAP has been suggested as an effective therapy to reduce psychosocial barriers and help individuals return to life roles including readiness to return to work. PGAP has been shown to be effective with some chronic health conditions however has not been specifically studied in mental health populations. The study consists of 10 one hour weekly therapy sessions that focus on reducing psychosocial risk factors that result in disability through the use of goal setting, activity planning and activation, monitoring and challenging thoughts about return to work, and problem solving. Participants will also be asked to complete short self-report questionnaires as well as a semi-structured interview about the participants anxiety, mood, impact of disability, and current functioning at the beginning of session one and within two weeks after session 10. Two short questionnaires will also be completed at each session measuring the degree to which the participants daily life impacts and is affected by anxiety or mood symptoms.

DETAILED DESCRIPTION:
The purpose of the present study is to determine the effectiveness of the Progressive Goal Attainment Program (PGAP) with individuals with anxiety and mood disorders. PGAP has been suggested as an effective therapy to reduce psychosocial barriers and help individuals return to life roles including readiness to return to work. PGAP has been shown to be effective with some chronic health conditions however has not been specifically studied in mental health populations.

The study consists of 10 one hour weekly therapy sessions with a clinician and follow the PGAP manual. The therapy sessions focus on reducing psychosocial risk factors that result in disability through the use of goal setting, activity planning, activation and re-engagement in activities, monitoring and challenging thoughts about return to work, and problem solving. Participants are also encouraged to participate in homework which involves daily activity planning, participating in planned activities, and tracking the activities completed. Participants will also be asked to complete short self-report questionnaires as well as a semi-structured interview about the participants anxiety, mood, impact of disability, and current functioning at the beginning of session one and within two weeks after session 10. Two short questionnaires will also be completed at each session measuring the degree to which the participants daily life impacts and is affected by anxiety or mood symptoms.

Our first hypothesis is that participants who receive PGAP will report significant reductions in functional disability as measured by self-report as well as by interview, decreases in self-reported work avoidance, increases in work readiness, and decreases in self-reported symptoms of anxiety and depression. Our second hypothesis is that mean reductions in the above-noted outcome variables will be similar in magnitude to those reported in published studies that have examined PGAP in chronic medically ill populations. Retention rates and satisfaction of the therapy will also be assessed to determine feasibility of implementing the program on a larger scale.

To examine the effectiveness of PGAP with participants with an anxiety or a mood disorder, the investigators will conduct a series of dependent sample t-tests on the outcome variables pre and post intervention. The investigators will also compare mean changes on the outcome variables to those in the published literature. The investigators will calculate retention rates with the aim of retaining more than 75% of participants, which is comparable to retention and drop out rates for psychotherapy trials with participants completing at least 8 out of 10 sessions or having returned to employment. Feasibility will also be measured by looking at satisfaction ratings. A minimal standard will be an average satisfaction rating across participants of midpoint (neutral) or above in terms of the therapy received.

ELIGIBILITY:
Inclusion Criteria:

Participants will be

1. between the ages of 18 and 65 years
2. have a principle diagnosis of an anxiety or mood disorder
3. have had changes in their work functioning, either currently not working due to their disability or on modified/reduced work.
4. be registered outpatients of the Anxiety Treatment and Research Clinic or Outpatient Mood Disorders Program, St. Joseph's Healthcare Hamilton,
5. are interested in return to work or have work related goals.

Exclusion Criteria:

1. current significant substance use
2. acute mental health (e.g. suicidality, psychosis, mania) that would interfere with the program completion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Impact of PGAP on disability (participant perception) | one year
  Level of disability will be measured using a modified version of the Pain Disability Index ( a 7 item self-report measure).

SECONDARY OUTCOMES:
Impact of PGAP on symptom change | one year
  Mood and anxiety symptoms will be measured using the Depression and Anxiety Stress Scales (a 21 item self-report measure).
Impact of PGAP on level of interference from mood and anxiety symptoms | one year
  Level of interference from mood and anxiety symptoms will be measured using the Illness Intrusiveness Rating Scale (13 item self-report measure).
Impact of PGAP on fear avoidance beliefs | one year
  Fear avoidance beliefs will be measured using the Fear Avoidance Beliefs Questionnaire (11 item self-report measure).
PGAP retention rates | one year
  Retention rates will be measured by tracking drop out rates.
Satisfaction with the PGAP | one year
  Satisfaction with the therapy will be assessed by using The Satisfaction with Therapy and Therapist Scale-Revised (13 item self-report measure).
Impact of PGAP on disability (clinician report) | one year
  Level of disability will be measured using the Multidimensional Scale of Independent Functioning (semi-structured interview).
Impact of PGAP on role functioning | one year
  Role functioning will be measured using the Multidimensional Scale of Independent Functioning (semi-structured interview).

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Colonerus, MADS, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No